CLINICAL TRIAL: NCT05860088
Title: The Effect of Beta-Alanine and Carnosine From Beef Intake on Muscle Fatigue in Older Adults
Brief Title: The Impact of Beef on Muscle Fatigue in Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Cydne Perry, Assistant Professor Applied Health Sciences, Indiana University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 14941
Record Dates: First submitted 2023-04-25; First posted 2023-05-16 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Muscle Weakness; Muscle; Fatigue, Heart; Older Adults
Keywords: Body Composition; Older Adults; Diet; Vegetarian; Meat; Beef; Controlled Feeding; Intervention
MeSH Terms: conditions — Muscle Weakness; Fatigue | interventions — Diet, Vegetarian

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beef Diet (Experimental): Participants will be randomized to consume the beef diet for 8 weeks. After a 2-week period, participants will cross-over to consume the vegetarian diet for 8 weeks.
  Interventions: Other: Beef Diet
- Vegetarian Diet (Experimental): Participants will be randomized to consume the vegetarian diet for 8 weeks. After a 2-week period, participants will cross-over to consume the beef diet for 8 weeks.
  Interventions: Other: Vegetarian Diet

INTERVENTIONS:
Other: Beef Diet — Controlled-Feeding Diet Intervention
  Arms: Beef Diet
Other: Vegetarian Diet — Controlled-Feeding Diet Intervention
  Arms: Vegetarian Diet

SUMMARY:
The goal of this controlled-feeding cross-over diet intervention is to compare a beef diet to a vegetarian diet on muscle fatigue in older adults. The aims are:

AIM 1: To test the hypothesis that muscle fatigue is attenuated in older adults consuming beef compared to older adults consuming a plant-based diet.

AIM2: To test the hypothesis that daily beef consumption improves biochemical indicators related to muscle fatigue.

Participants will be randomized to consume either a beef-based diet or vegetarian diet under controlled-feeding conditions for 8 weeks. After a 2-week washout period, participants will cross-over to consume either the beef diet or vegetarian diet for 8 weeks. Body composition and functional muscle outcomes will be measured during each 8-week feeding period. Blood samples will also be collected.

ELIGIBILITY:
Inclusion Criteria

* Ages 60-85 years
* Ability to eat study diet meals for a total of 16 weeks
* Ability to perform sit-to-stand chair and 6-minute walking tests based on results from PAR-Q questionnaire
* Ability to provide fasted blood samples
* Access to transportation
* Willing to abstain from alcohol consumption and/or use illicit drug use for each 8-week intervention period
* Ability to consent to participating in this study
* English-speaking
* Body mass index between 18.5 (normal) and 39.9 (obese) kg/m2
* Minimum total body weight of 110 pounds
* Non-anemia hemoglobin values: Females - >12.0 grams/dL; Men - >13.0 grams/dL
* Able to ambulate without assistance
* Physician's clearance for study participation (required prior to baseline testing)

Exclusion Criteria

* Inability or refusal to sign the informed consent
* Significant orthopedic limitations or other contraindications to exercise
* Inability or refusal to perform muscle fatigue tests
* Has dietary restrictions that prevent to consumption of beef, soy and/or wheat
* Has liver or kidney complications
* Live or work >25 miles from Bloomington study site or does not have transportation to the study site
* Anticipate elective surgery during the study period
* Diagnosis of progressive neurological disorders, musculoskeletal disorders, osteoarthritis, rheumatoid arthritis
* Fracture or serious injury in the last 6 months
* Stroke, revascularization, deep vein thrombosis, or pulmonary embolism in the past 12 months
* Severe cardiovascular disease, uncontrolled systemic hypertension, chronic pulmonary disease
* Plan to move residence or travel out of the local area during the study period
* Current use of anti-coagulants (e.g. Coumadin or Warfarin)
* Current use of prescription medications that affect heart rate or blood vessel dilation
* Psychological or social characteristics that would interfere with their ability to fully participate in the study

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-07-10 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change in Sit-to-Stand Chair Test | Weeks 0, 4, 8
  The change in muscle strength observed in each diet condition will be evaluated through the Sit-To-Stand Chair Test. The number of times a participant comes to a full standing position (from a seated position) in 60 seconds will be recorded.
Change in 6-minute walk | Weeks 0, 4, 8
  The change in muscle strength observed in each diet condition will be evaluated through the 6-Minute-Walk-Test. The distance walked by a participant during the 6 minute test period will be recorded.
Retention of Participants | Through study completion, approximately 16 weeks
  The percentage of randomized participants completing the 16-week diet intervention trial.
Adherence to Study Diets | Through study completion, approximately 16 weeks
  Participant adherence to the study diets will be evaluated.

SECONDARY OUTCOMES:
Change in Lactate | Weeks 0, 4, 8
  Measures of muscle fatigue will be evaluated through blood biomarkers.
Change in Beta-Alanine | Weeks 0, 4, 8
  Measures of muscle fatigue will be evaluated through blood biomarkers.
Change in Carnosine | Weeks 0, 4, 8
  Measures of muscle fatigue will be evaluated through blood biomarkers.
Change in Amino Acids | Weeks 0, 4, 8
  Measures of muscle fatigue will be evaluated through blood biomarkers.

CONTACTS AND LOCATIONS:
Overall Officials: Cydne A Perry, PhD, Principal Investigator — Indiana University, Bloomington
Locations (1):
- Indiana University Bloomington, Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: No